CLINICAL TRIAL: NCT03868098
Title: A Randomized, Double-Blind, Intra-Individual, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of Different Application Rates of Topically Applied Crisaborole Ointment 2% in Adult Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: Different Application Rates of Crisaborole Ointment 2% in Adults With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6049
Record Dates: First submitted 2019-03-07; First posted 2019-03-08 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Intervention Model Description: Intra-individual
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisaborole 2% (application rate A, B, C) (Active Comparator): Crisaborole (Marketed drug)
  Interventions: Drug: Crisaborole 2%
- Placebo ointment (vehicle) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Crisaborole 2% — Crisaborole ointment 2% (application rate A, B, C) for 15 days (double blind)
  Other Names: Eucrisa
  Arms: Crisaborole 2% (application rate A, B, C)
Drug: Placebo ointment — Placebo ointment (vehicle)
  Arms: Placebo ointment (vehicle)

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of 3 different application rates of topically applied Crisaborole ointment 2% over vehicle in adults with mild to moderate atopic dermatitis (AD). In each subject four application areas will be identified. Each subject will receive 4 treatments: the 3 different application rates of the active treatment and the vehicle. The areas will be randomly assigned to treatment with topical Crisaborole ointment 2% and vehicle, once daily, for 2 weeks, without occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of active atopic dermatitis (AD) with at least 6 month history prior to screening and that has been clinically stable for 1 month.
* Has four application areas of 3 cm in diameter with a TSS of ≥5 and TAA of moderate at Day 1. The application areas must not be located on the face, scalp, axillae, groin, genitals, hands, and feet. The application areas should be ≥1 cm apart.

Exclusion Criteria:

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has clinically infected AD.
* Subject has a Fitzpatrick's Skin Phototype ≥5.
* Subject is known to have immune deficiency or is immunocompromised.
* Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Subjects with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or successfully treated localized carcinoma in situ of the cervix are not to be excluded.
* Subject had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* Subject has any clinically significant medical condition that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
* Subject has a known history of chronic infectious disease (eg, hepatitis B, hepatitis C, or infection with human immunodeficiency virus).
* Subject with a known lack of efficacy to crisaborole.
* Subject has a known or suspected allergy to crisaborole, including any non-medicinal ingredient, or component of the container.
* Subject has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Total Signs Score (TSS) | Baseline, Day 15
  Change from baseline in TSS in target lesions treated with crisaborole ointment 2% or vehicle at Day 15.
  Total Signs Score (TSS) of the lesion is the assessment of the severity of erythema, edema/papulation, excoriation, and lichenification. Each of these subscales is scored independently using the 4-point severity scale with a value range from 0 to 3; 0 is the minimum (best) and 3 is the maximum (worst). The total score is computed by the sum of each subscale where the total ranges from the minimum 0 (best) to the maximum 12 (worst).

SECONDARY OUTCOMES:
Total Signs Score (TSS) | Baseline, Day 8, Day 15
  Change from baseline in lesion severity as measured by TSS at Day 8 and Day 15
  Total Signs Score (TSS) of the lesion is the assessment of the severity of erythema, edema/papulation, excoriation, and lichenification. Each of these subscales is scored independently using the 4-point severity scale with a value range from 0 to 3; 0 is the minimum (best) and 3 is the maximum (worst). The total score is computed by the sum of each subscale where the total ranges from the minimum 0 (best) to the maximum 12 (worst).
Target Area Assessment (TAA) | Change from baseline in TAA at Day 8 and Day 15.
  Change from baseline in TAA at Day 8 and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Medical Director
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No